CLINICAL TRIAL: NCT05896397
Title: European Aortic Data Collection Project
Acronym: EADC
Status: Recruiting | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: MDR-2091
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Complex Abdominal Aortic Aneurysm; Thoracoabdominal Aortic Aneurysm; Aortic Arch Aneurysm; Chronic Aortic Dissection
Keywords: Complex aortic repair; Aortic aneurysm; Aortic dissection; Fenestrated/branched endograft; Custom-made endovascular graft
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aneurysm, Aortic Arch; Aortic Aneurysm; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endovascular Aortic Treatments — Use of Cook's custom-made endovascular grafts to treat complex abdominal, thoracoabdominal aortic diseases, or aortic arch diseases such as aneurysms and dissections.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of Cook's various Custom-Made Stent-graft Devices (CMD) used for endovascular treatment of the aorta and related diseases by collecting information on the real-world use of the devices.

The study results will be used to support the continuation of the CMDs on the market. In addition, the study will support the manufacturers obligation for post market product surveillance as well as Cook's technology development.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will be treated with a Cook CMD

Exclusion Criteria:

1. Patients who declare they are unable to complete clinical follow-up visit at the time of enrollment, or
2. Patients or his/her legally authorized representative objects to extraction of patient's data from the medical record, or unwilling to sign the Informed Consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving a Cook custom made endovascular graft within the scope of the study in a maximum of 20 clinical sites in Europe.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Rate of treatment success | 12 months
  Procedural treatment success is defined as successful access to the arterial system using remote arterial exposure, percutaneous technique or open surgical conduits. Success is also defined as successful delivery and deployment of the aortic graft and all stent components, side branch catheterization and placement of bridging stents and patency of all aortic modular stent graft components and intended side branch components.
Rate of safety outcomes | 30 days
  Safety outcomes is defined as freedom from major adverse events (all-cause mortality, myocardial infarction, disabling stroke, renal failure requiring new-onset dialysis, respiratory failure requiring prolonged (>24hrs) mechanical ventilation or reintubation, paraplegia, bowel ischemia requiring surgical resection or not resolving with medical therapy)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Haulon, MD,PhD, Principal Investigator — Hopital Marie Lannelongue
Locations (18):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (2):
  - Hopital Marie Lannelongue, Le Plessis-Robinson
  - CHU de Lille, Lille
- Germany (4):
  - University Hospital Hamburg Eppendorf, Hamburg
  - LMU Klinikum Munich, Munich
  - St. Franzikus-Hospital Munster, Münster
  - Klinnikum Nurnberg, Nuremberg
- Italy (4):
  - PoliclinicoS Orsola Malpighi, Bologna
  - Orsola Maplighi, Bologna
  - Ospedal Policlinico San Martino-HSM, Genova
  - IRCCS San Raffaele Hospital, Milan
- Sweden (2):
  - Skane University Hospital Malmo, Malmo
  - Uppsala University Hospital, Uppsala
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - North Bristol NHS Trust, Bristol
  - St Thomas' Hospital, London
  - St Barthowlomew's, London

IPD SHARING:
Plan to Share IPD: Undecided